CLINICAL TRIAL: NCT00308178
Title: Dose Dense AB1-007 (Abraxane) in Adjuvant Chemotherapy for Breast Cancer: A Feasibility Study
Brief Title: Dose Dense Abraxane in Adjuvant Chemotherapy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harold J. Burstein, MD, PhD (Other)
Collaborators: Celgene Corporation (Industry); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Harold J. Burstein, MD, PhD, Associate Professor of Medicine, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-249
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: Abraxane; dose-dense chemotherapy; taxol
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: Abraxane — Following 4 cycles (8 weeks) of adjuvant chemotherapy (adriamycin and cytoxan), abraxane will be give every 2 weeks for 4 cycles(8 weeks)

SUMMARY:
The purpose of this trial is to see if Abraxane, which is a new form of paclitaxel, is safe as a replacement form of paclitaxel in dose-dense chemotherapy. This trial will also determine if using Abraxane will allow patients to receive treatment every two weeks without requiring injects of G-CSF, a white blood cell stimulating growth factor.

DETAILED DESCRIPTION:
* Patients will receive regular chemotherapy every 2 weeks for up to 8 cycles (approximately 16 weeks total)of treatment. During the first four cycles patients will be treated with Adriamycin and Cytoxan, and for the second four cycles they will be treated with Abraxane.
* Patients will be taught to give themselves injections with either short or long acting G-CSF as prescribed by their doctor for the first four cycles of chemotherapy. During the last four cycles (while the patient is taking Abraxane) they will not receive G-CSF unless they have low blood counts.
* If the patient has HER-2 positive breast cancer, they will also receive 52 weeks of Herceptin as part of standard cancer care and will begin to receive Herceptin at the same time they begin Abraxane (after 4 cycles of adriamycin and cytoxan treatment).
* This study involves a series of Quality of Life Questionnaires that will be completed prior to beginning study treatment, then again at 2 months, 4 months, 6 months, and 1 year after starting study treatment.
* The following tests and procedures will be performed at the time periods specified. Cycle 1-4 Day 1: Physical exam, vital signs, and blood tests. Cycle 5 Day 1: Physical exam, vital signs, blood tests, RVG (measurement of heart function) and questionnaire. Cycle 6 & 7 Day 1: Physical exam, vital signs, and blood tests. Cycle 8 Day 1: physical exam, vital signs, blood tests, questionnaire. Follow-up (6 months and 1 year after cycle 1 day 1): questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer, with clinical stage I, II, or III disease
* Must register at the beginning of adjuvant or neoadjuvant chemotherapy
* 18 years of age or older
* ECOG performance status of 0 or 1
* Normal organ and marrow function

Exclusion Criteria:

* Previous cytotoxic chemotherapy or therapeutic radiation therapy for any reason
* Pregnant or nursing
* Receiving any other investigational agents
* Patients with Stage IV breast cancer
* Current grade II or greater peripheral neuropathy or prior history of grade II or greater neuropathy
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Immune deficiency when treated with marrow-suppressive therapy or HIV-positive patients receiving anti-retroviral therapy
* Patients with sickle cell disease
* Known history of hyperviscosity syndrome
* Patients on lithium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-03; Primary Completion 2006-09 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility and toxicity of Abraxane after chemotherapy as part of dose-dense adjuvant chemotherapy for breast cancer. | 2 years

SECONDARY OUTCOMES:
To evaluate the feasibility of administering Abraxane on a dose dense schedule without G-CSF support | 2 years
to estimate the percentage of patients with various grades of hematologic toxicity, neurotoxicity, and other non-hematologic toxicity associated with dose-dense Abraxane | 2 years
to evaluate quality of life. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Harold Burstein, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massacusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts